CLINICAL TRIAL: NCT03962491
Title: Using Mobile-based Contingency Management to Promote Daily Self-monitoring of Pain Severity and Prescription Opioid Use in a Primary Care Sample of Chronic Pain Patients
Brief Title: Mobile-Based Contingency Management to Promote Daily Self-monitoring in Primary Care Patients
Acronym: ProMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20013828; 1R36DA046671 (NIH)
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Self-Monitoring Surveys (Other): Asked to complete daily self-monitoring surveys.
  Interventions: Behavioral: Daily Self-Monitoring Surveys
- Daily Self-Monitoring Surveys + Contingency Management (Experimental): Asked to complete daily self-monitoring surveys, with opportunity for monetary rewards.
  Interventions: Behavioral: Daily Self-Monitoring Surveys + Contingency Management

INTERVENTIONS:
Behavioral: Daily Self-Monitoring Surveys + Contingency Management — Asked to complete a brief (5-minute) survey with questions related to pain experience and related measures every day for 28 days using the DynamiCare smartphone app, with the opportunity for monetary rewards for completing daily surveys.
  Arms: Daily Self-Monitoring Surveys + Contingency Management
Behavioral: Daily Self-Monitoring Surveys — Asked to complete a brief (5-minute) survey with questions related to pain experience and related measures every day for 28 days using the DynamiCare smartphone app.
  Arms: Daily Self-Monitoring Surveys

SUMMARY:
This project examines the efficacy and feasibility of contingency management (CM), delivered using a novel, fully automated CM app (DynamiCare Rewards), to promote daily self-monitoring of pain symptom severity and related variables (e.g., mood, sleep), as well as Rx opioid, alcohol, marijuana, cannabidiol (CBD), and Rx benzodiazepine use in a sample of chronic pain patients. The project will conduct a 2-arm randomized clinical trial (RCT) comparing those receiving reinforcement escalating with continuous performance of the target behavior (CM group) vs those asked to complete the survey but will not be incentivized (C group).

DETAILED DESCRIPTION:
Prescription (Rx) opioid misuse is a significant public health problem and the CDC has declared an opioid epidemic (Dowell, Haegerich, & Chou, 2016). Chronic pain patients, often prescribed opioids for pain management, represent a particularly vulnerable population (e.g., Boscarino et al., 2011). Responsible opioid prescribing depends on effective identification of misuse and comprehensive understanding of pain-related variables (Dowell, Haegerich, & Chou, 2016). Self-report tracking via smartphone apps is a promising solution, but difficulties with adherence have been found to impede the use of remote self-monitoring among chronic pain patients (e.g., Jamison et al., 2016), even with the inclusion of non-monetary rewards (Jamison et al., 2017). One robust strategy for improving adherence is contingency management (CM). While CM has been widely used in research, the translation to clinical practice has met with resistance due, in large part, to practical barriers (e.g., Carroll, 2014).

As a Stage 1 behavioral therapies development project (Rounsaville et al., 2001), the goal of this study is to examine the efficacy and feasibility of CM, delivered using a novel, fully automated CM app (DynamiCare), to promote daily self-monitoring of pain symptom severity and related variables (e.g., mood, sleep), as well as Rx opioid, alcohol, marijuana, cannabidiol (CBD), and Rx benzodiazepine use in a sample of chronic pain patients. The target behavior will be objectively defined as completing daily self-monitoring surveys via the app for which those randomized to CM will earn incentives.

Participants will complete baseline assessment, followed by random assignment to either the experimental (CM) or control (C) group. All participants will then download the app onto their smartphone and be provided with instruction in its use. Based on the work by Petry et al. (2005) and Olmstead and Petry (2009), the CM group will receive reinforcement escalating with continuous performance of the target behavior while the C group will be asked to complete the survey, but will not receive incentivizes. Both groups will receive reminders to complete the daily survey. Follow-up assessments (including behavioral and psychological measures) will occur at intervention completion (28-days post-randomization) and both CM and C group members will be compensated for their time and effort.

The specific aims of this project are to: 1) Compare number of completed daily self-monitoring surveys in CM and C groups; 2) Compare longest sustained period of daily survey completion in CM and C groups; 3) Examine agreement between daily survey and 28-day follow-up visit reports of Rx opioid, alcohol, marijuana, cannabidiol (CBD), and Rx benzodiazepine use in CM and C groups; 4) Examine feasibility and acceptability of CM app implementation targeting self-monitoring of pain severity, related factors, and Rx opioid, alcohol, marijuana, cannabidiol (CBD), and Rx benzodiazepine use; and 5) Estimate effect-size to be used to perform power analyses and sample size calculations as part of the design of a larger RCT.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age;
2. own a study-compatible smartphone (iPhone or Android device);
3. report non-cancer related chronic pain (consistent daily pain) for 3 months or greater;
4. able to provide informed consent for study participation;
5. used prescription opioids in the past 30 days; and
6. having ever been prescribed 1 or more opioid medication(s) for pain management.

Exclusion Criteria:

1. currently pregnant;
2. presenting with language barriers, cognitive impairment, or serious medical or psychiatric illness that in the opinion of the Investigator would preclude them from providing informed consent or participating in the study; and
3. visual impairment or motor impairment that would interfere with use of a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dace Svikis, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Self-Monitoring Surveys | Daily Self-Monitoring Surveys + Contingency Management
Started | 35 | 46
Completed | 31 | 41
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Self-Monitoring Surveys | Daily Self-Monitoring Surveys + Contingency Management | Total
Number analyzed (Participants) | 35 | 46 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.71 (12.39) | 44.02 (16.12) | 44.76 (14.55)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 28 | 33 | 61
  Male | 7 | 12 | 19
  Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 32 | 40 | 72
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 32 | 40 | 72
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Number; unit: participants]
  United States | 35 | 46 | 81

OUTCOME MEASURES:

1. Primary Outcome: Number of Daily Self-monitoring Surveys Completed
Description: Number of days daily surveys completed
Time Frame: 28-day daily survey period
Measure: Mean (Standard Deviation); unit: Surveys completed
Arm/Group | Daily Self-Monitoring Surveys | Daily Self-Monitoring Surveys + Contingency Management
Number analyzed (Participants) | 35 | 46
Surveys completed | 23.06 (6.97) | 26.09 (3.85)

2. Primary Outcome: Longest Period of Sustained Adherence to Daily Survey Completion
Description: Largest number of consecutive days wherein daily surveys were completed
Time Frame: 28-day daily survey period
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Daily Self-Monitoring Surveys | Daily Self-Monitoring Surveys + Contingency Management
Number analyzed (Participants) | 35 | 46
number of days | 17.11 (9.36) | 22.07 (7.76)

3. Secondary Outcome: Daily Survey Completion Time
Description: Mean time to complete daily surveys
Time Frame: 28-day daily survey period
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Daily Self-Monitoring Surveys | Daily Self-Monitoring Surveys + Contingency Management
Number analyzed (Participants) | 35 | 46
minutes | 8.71 (33.03) | 5.78 (9.66)

4. Secondary Outcome: CM App Acceptability
Description: CM App Acceptability was measured using a 8 item scale asking about experiences using the app. Each item was rated on a 0 - 10 Likert scale with higher scores indicating more positive responses. Scores for each item are reported separately.
Time Frame: 28-day follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Daily Self-Monitoring Surveys | Daily Self-Monitoring Surveys + Contingency Management
Number analyzed (Participants) | 35 | 46
score on a scale
  Easy to use | 7.71 (1.11) | 6.67 (1.23)
  Overall satisfaction | 7.78 (1.48) | 7.31 (1.49)
  Useful | 6.58 (2.17) | 6.82 (2.30)
  Appealing | 7.13 (2.03) | 7.50 (1.69)
  Bothersome | 6.95 (2.16) | 5.50 (3.04)
  Willing to use | 7.09 (2.43) | 8.11 (1.05)
  Help you cope with pain | 4.25 (2.15) | 4.87 (2.45)

5. Other Pre Specified Outcome: Agreement Between Daily Survey and 28-day Follow-up Reports of Alcohol Use
Time Frame: 28-day daily survey period to 28-day follow-up
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Agreement Between Daily Survey and 28-day Follow-up Reports of Rx Opioid Use
Time Frame: 28-day daily survey period to 28-day follow-up
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Agreement Between Daily Survey and 28-day Follow-up Reports of Rx Benzodiazepine Use
Time Frame: 28-day daily survey period to 28-day follow-up
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Agreement Between Daily Survey and 28-day Follow-up Reports of Marijuana Use
Time Frame: 28-day daily survey period to 28-day follow-up
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Agreement Between Daily Survey and 28-day Follow-up Reports of Cannabidiol Use
Time Frame: 28-day daily survey period to 28-day follow-up
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: None - adverse event data was not collected
Description: Adverse event data was not collected.
Arm/Group | Daily Self-Monitoring Surveys | Daily Self-Monitoring Surveys + Contingency Management
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03962491/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03962491/ICF_001.pdf